CLINICAL TRIAL: NCT04412720
Title: Effects of Aerobic and Respiratory Exercises on Asthma Clinical Control
Brief Title: Aerobic and Respiratory Exercises on Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2491900
Record Dates: First submitted 2020-05-21; First posted 2020-06-02 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2020-01

CONDITIONS: Asthma
Keywords: Aerobic exercises; Respiratory exercises; Asthma clinical control
MeSH Terms: conditions — Asthma | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All the measurements will be performed by a professional blinded to the groups. The same assessor will be maintained to perform the evaluations before and after the intervention. The professionals involved with the evaluations will be different from the professionals involved on the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic and Breathing Exercises (Experimental): The experimental intervention will be aerobic and breathing exercises.
  Interventions: Other: Aerobic and Breathing Exercises
- Aerobic and Stretching Exercises (Active Comparator): The active comparative intervention will be aerobic and stretching exercises.
  Interventions: Other: Aerobic and Stretching Exercises

INTERVENTIONS:
Other: Aerobic and Breathing Exercises — Aerobic exercises will be performed on a treadmill, twice a week, totaling 20 sessions of 60 minutes each. The initial intensity will be 50% to 60% of maximum heart rate and the progression will take place according to the level of effort (Borg) in the last two sessions. In addition, following the aerobic training, Buteyko Breathing Technique also will be performed during 20 minutes each exercise, in the same treatment session. During the first two weeks, the patient will learn the technique supervised by a physical therapist. In addition, the patients will receive a breathing exercise booklet for in-home training. Before and after each session, patients will be evaluated in relation to blood pressure, heart rate, oxygen saturation and asthma symptoms.
  Arms: Aerobic and Breathing Exercises
Other: Aerobic and Stretching Exercises — Aerobic exercises will be performed on a treadmill, twice a week, totaling 20 sessions of 60 minutes each. The initial intensity will be 50% to 60% of maximum heart rate and the progression will take place according to the level of effort (Borg) in the last two sessions. In addition, following the aerobic training, stretching exercises will be performing for major muscle groups, during 30 seconds each one. The patients will receive a stretching exercise booklet for in-home training.
  Arms: Aerobic and Stretching Exercises

SUMMARY:
Many studies have reported the benefits of aerobic and breathing exercises such as, reduction of symptoms and reduced the use of medications, the number of crises, exercise induced bronchoconstriction (EIB), and improvement in health-related quality of life (HRQoL). This study will be a randomized and controlled trial (RCT) with 2 parallel arms and blinded assessment. Fifty-four moderate or severe patients with asthma under optimized medication will be randomly assigned (computer-generated) into either aerobic+breathing exercises (AB) or aerobic+stretching exercises (AS). All patients will receive the same educational session and will perform the physical exercise proposed for the group for 12 weeks, 2 times/week, 60-minute sessions; however, the AB group will perform Buteyko breathing technique and AS will perform muscle stretching exercise. All patients will be assessed to clinical control, quality of life, psychosocial symptoms, pulmonary function, functional capacity, physical activity levels, sleep quality, thoracoabdominal mechanics, hyperventilation symptoms, and asthma exacerbation. The data normality will be analyzed by Kolmogorov-Smirnov. The variables obtained before interventions will be compared using the t-test or Mann-Whitney U-test. Comparisons of the outcomes initial and final data will be analyzed with repeated measures ANOVA with appropriate post hoc test. The significance level will be set to 5% for all tests.

DETAILED DESCRIPTION:
Many studies have reported the benefits of aerobic and breathing exercises such as, reduction of symptoms and reduced the use of medications, the number of crises, exercise induced bronchoconstriction (EIB), and improvement in health-related quality of life (HRQoL). This study will be a randomized and controlled trial (RCT) with 2 parallel arms and blinded assessment. Fifty-four moderate or severe patients with asthma under optimized medication will be randomly assigned (computer-generated) into either aerobic+breathing exercises (AB) or aerobic+stretching exercises (AS). All patients will receive the same educational session and will perform the physical exercise proposed for the group for 12 weeks, 2 times/week, 60-minute sessions; however, the AB group will perform Buteyko breathing technique and AS will perform muscle stretching exercise. All patients will be assessed to clinical control, quality of life, psychosocial symptoms, pulmonary function, functional capacity, physical activity levels, sleep quality, thoracoabdominal mechanics, hyperventilation symptoms, and asthma exacerbation. The data normality will be analyzed by Kolmogorov-Smirnov. The variables obtained before interventions will be compared using the t-test or Mann-Whitney U-test. Comparisons of the outcomes initial and final data will be analyzed with repeated measures ANOVA with appropriate post hoc test. The significance level will be set to 5% for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Asthma moderate and severe with diagnosed according to the Global Initiative for Asthma (GINA) 2020
* Sedentary (< 150 min of moderate to vigorous physical activity/week)
* Body Mass Index ≥18.5 kg/m2 and <35 kg/m2
* Medical treatment, for at least 6 months
* Clinically stable (i.e., no exacerbation or changes in medication for at least 30 days)

Exclusion Criteria:

* Cardiovascular, musculoskeletal or other chronic lung diseases
* Active Cancer
* Pregnant
* Uncontrolled hypertension or diabetes
* Current smoker or ex smoker (>10 pack-years)
* Psychiatric disease or cognitive deficit

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in asthma clinical control | Change from baseline to 10 weeks of intervention
  Clinical control will be evaluated by the Asthma Control Questionnaire (ACQ). The ACQ contains 7 items rated on a 7-point scale (0 = without limitation, 6 = maximum limitation), with a higher score indicating worse control. Scores lower than 0.75 are associated with good asthma control, whereas scores greater than 1.5 are indicative of poorly controlled asthma, and a change of at least 0.5 points in the ACQ score is regarded as clinically significant.

SECONDARY OUTCOMES:
Change in health related quality of life | Change from baseline to 10 weeks of intervention
  Health related quality of life will be assessed by Asthma Quality Life Questionnaire (AQLQ). The AQLQ consists of 32 items rated on a 7-point scale (1 = great deal, 7 = not at all) divided into the following 4 domains: activity limitations, symptoms, emotional function and environmental stimuli. Higher AQLQ scores indicate a better quality of life, and treatments resulting in a 0.5-point increase in scores following an intervention are considered to be clinically effective.
Change in psychosocial symptoms | Change from baseline to 10 weeks of intervention
  Symptoms of anxiety and depression symptoms will be assessed by the Hospital Anxiety and Depression scale (HADs), which consists of 14 items divided into 2 subscales (7 for anxiety and 7 for depression). Each item is scored from 0 to 3, with a maximum score of 21 points for each subscale. A score greater than 8/9 in each subscale suggests a diagnosis of either anxiety and/or depression.
Change in pulmonary function in absolute values | Change from baseline to 10 weeks of intervention
  Lung volumes will be assessed by Spirometry. The variables which will be assessed are Forced Vital Capacity (FVC) and Forced Expiratory Volume in first 1 second (FEV1), all them in liters.
Change in pulmonary function in predict values | Change from baseline to 10 weeks of intervention
  The variables which will be assessed are predicted values for brazilian population of Forced Vital Capacity (FVC), Forced Expiratory Volume in first 1 second (FEV1), and FEV1/FVC ratio.
Change in functional capacity | Change from baseline to 10 weeks of intervention
  The functional capacity will be assessed by the Incremental Shuttle Walking Test (ISWT)
Change in physical activity levels | Change from baseline to 10 weeks of intervention
  Physical activity and sedentary behaviour will be objectively quantified using a movement sensor (ActiGraph, Pensacola, USA) for 7 consecutive days on the hip using an elastic belt. Sedentary behaviour will be quantify by the time spent sedentary (< 100 counts/min).
Change in sleep quality | Change from baseline to 10 weeks of intervention
  Sleep quality will be objectively quantified using a movement sensor (ActiGraph, Pensacola, USA) for 7 consecutive nights on the wrist (non-dominant side), and by Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 9 items divided into the following 7 domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. A global sum of "5"or greater indicates a "poor" sleeper.
Change in thoracoabdominal mechanics | Change from baseline to 10 weeks of intervention
  The thoracoabdominal mechanics will be assessed by optoelectronic plethysmography
Change in hyperventilation symptoms | Change from baseline to 10 weeks of intervention
  Hyperventilation symptoms will be assessed by the Nijmegen Questionnaire which consists of 16 items. Each item is scored from 0 to 4. A score greater than 23 suggest a positive diagnosis of hyperventilation.
  syndrome.
Change in asthma exacerbation | Change from baseline to 10 weeks of intervention
  Asthma exacerbation will be assessed by the following criteria: the use of ≥4 puffs of rescue medication per 24 hours during a 48-hour period, a need for systemic corticosteroids, an unscheduled medical appointment, and either a visit to an emergency room or hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Study Director — University of Sao Paulo General Hospital
Locations (1):
- Celso Ricardo Fernandes de Carvalho, São Paulo, Brazil